CLINICAL TRIAL: NCT05933239
Title: A Phase II Study to Evaluate the Imaging Potential of 68GaNOTA-Anti-MMR VHH2 for in Vivo Imaging of MMR-expressing Macrophages by Means of Positron Emission Tomography (PET) in Patients With Non-small Cell Lung Cancer (NSCLC)
Brief Title: Macrophage Imaging Using Ga-MMR-VHH2 in Lung Cancer Patients
Acronym: MAGMA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UZBRU_VHH2_4
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: PET/CT; MMR-PET/CT; Macrophage PET/CT; CD206
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients diagnosed with non-small cell lung cancer (NSCLC), planned for standard-of-care surgery (Other)
  Interventions: Drug: 68GaNOTA-Anti-MMR-VHH2

INTERVENTIONS:
Drug: 68GaNOTA-Anti-MMR-VHH2 — Injection of the radiopharmaceutical and PET/CT imaging

SUMMARY:
Phase II study to evaluate the clinical potential of 68GaNOTA-anti-MMR-VHH2 for in vivo imaging of Macrophage Mannose Receptor (MMR)-expressing Macrophages by means of Positron Emission Tomography (PET) in patients with non-small cell lung cancer (NSCLC) planned for surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given informed consent
* Patients at least 18 years old
* Patient with local, locally advanced or metastatic disease of non-small cell lung cancer, who is planned for resection or surgical biopsy of at least one lesion. In order to minimise partial volume effect, the diameter of the tumour to be resected or biopsied should be ≥ 10 mm in short axis for invaded adenopathies and ≥ 10 mm in long axis for all other types of lesions
* Patients who participated already in this study can be included if the subject meets all of the inclusion and none of the exclusion criteria at time of second inclusion.

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 3 or higher
* Pregnant patients
* Breast feeding patients
* Patients with any serious active infection
* Patients who have any other life-threatening illness or organ system dysfunction, which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the test radiopharmaceutical
* Patients who are unlikely to cooperate with the requirements of the study
* Patients who are unwilling and/or unable to give informed consent
* Patients at increased risk of death from a pre-existing concurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of uptake of 68GaNOTA-Anti-MMR-VHH2 in a NSCLC lesion before surgery with the immunohistological MMR-staining of the excised lesion. | Resection of lesion up to 21 days after PET/CT
  PET/CT and immunohistochemistry will be assessed using a (semi-)quantitative scale.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Lahoutte, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium